CLINICAL TRIAL: NCT07242378
Title: Evaluating Knowledge Mobilization Sustainability Approaches for Stress Management in University Students
Brief Title: Evaluating Knowledge Mobilization Sustainability Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor Emerita, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-05-100
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stress; Coping; Well-being; Mindfulness; Behaviour Change; Adherence; Digital Intervention
Keywords: stress management; maintenance of behaviour change; strategy use; self-guided resource; university students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Workshop Booster Sessions (Experimental): Two 45-minute online workshop booster sessions presented about two months apart, led by two trained undergraduate peer facilitators with 10 to 20 participants per session. Students were taught strategies to support their use of stress management techniques. Session themes included: (a) understanding values; (b) goal setting; (c) planning for challenges; (d) awareness of resources; (e) facing setbacks; (f) building a community of practice; and (g) general tips for getting started. Following each workshop session, students were emailed a brief one-page resource sheet with links to the strategies for habit formation presented in the session.
  Interventions: Behavioral: Sustainability of stress management strategy use; Behavioral: Stress management
- Experimental: Community Drop-in Sessions (Experimental): Five monthly 20-minute online community drop-in sessions held over a five-month period, led by the same peer facilitators as in the workshop and with 10-15 participants. These community drop-in sessions covered identical content to that of the workshop sessions, but were delivered in a more informal discussion format (i.e., no PowerPoint presentation). Students were taught strategies to support their use of stress management techniques. Session themes included: (a) understanding values; (b) goal setting; (c) planning for challenges; (d) awareness of resources; (e) facing setbacks; (f) building a community of practice; and (g) general tips for getting started. Following each community drop-in session, students were emailed a brief one-page resource sheet with links to the strategies for habit formation presented in the session.
  Interventions: Behavioral: Sustainability of stress management strategy use; Behavioral: Stress management
- Experimental: Infographic Reminders (Experimental): Ten brief digital infographic reminders (one to two pages each) emailed to students once every two weeks over a five-month period.The infographics including strategies with interactive links to support their use of stress management techniques. Session themes included: (a) understanding values; (b) goal setting; (c) planning for challenges; (d) awareness of resources; (e) facing setbacks; (f) building a community of practice; and (g) general tips for getting started.
  Interventions: Behavioral: Sustainability of stress management strategy use; Behavioral: Stress management
- No Sustainability Intervention: Inactive Control (Active Comparator): Participants in the inactive control group did not receive any sustainability support until the end of the study.
  Interventions: Behavioral: Stress management

INTERVENTIONS:
Behavioral: Sustainability of stress management strategy use — Then, different sustainability approaches (workshop boosters, community drop-ins, infographic reminders) were developed to ensure equivalent content across: (a) psychoeducation on habit formation and maintenance of behaviour change; and (b) embedded skills-based practice of habit formation. Themes addressed in the sustainability approaches included: (a) understanding values; (b) goal setting; (c) planning for challenges; (d) awareness of resources; (e) facing setbacks; (f) building a community of practice; and (g) general tips for getting started.
  Arms: Experimental: Community Drop-in Sessions; Experimental: Infographic Reminders; Experimental: Workshop Booster Sessions
Behavioral: Stress management — All groups received a digital infographic with interactive links with stress management strategies. Stress management strategies touched on 4 main areas which included (a) pause/break; (b) positive awareness; (c) kindness to self; and (d) social support.

SUMMARY:
The overarching objective of the current study is to evaluate the effectiveness, acceptability, strategy use, and maintenance of behaviour change of different stress management sustainability groups. Furthermore, the study aims to examine how these sustainability groups and maintenance of behaviour change may impact student wellness in the long term. Specifically, objective 1 sought to compare three commonly employed approaches for sustainability of stress management strategy use (workshop booster sessions, online community drop-ins, digital infographic reminders) and an inactive control group (no support) in terms of their (1.1) effectiveness on wellness outcomes (i.e., stress, healthy and unhealthy coping capacity, mindfulness, coping self-efficacy, and well-being), (1.2) acceptability, (1.3) strategy use, and (1.4) maintenance of behaviour change over time. It was hypothesized that the community drop-in sustainability group would have greater effectiveness, strategy use, and maintenance of behaviour change compared to the other sustainability groups and inactive control. This hypothesis aligns with the literature across both sustainability supports and maintenance of behaviour change-related indices, suggesting that social support is a key element to sustained strategy use (Borghouts et al., 2021; Kelders et al., 2012; Kwasnicka et al., 2016). No specific hypothesis was made for which sustainability approach would be rated as most (H1.2) acceptable given this is a novel area of research.

Objective 2 sought to examine (2.1) whether maintenance of behaviour change at post (T2) predicted wellness outcomes (i.e., stress, healthy and unhealthy coping capacity, mindfulness, coping self-efficacy, and well-being) at 6-month follow-up (T4), and whether this relationship was differentially moderated by sustainability group. It was hypothesized (H2.1) that maintenance of behaviour change at post would positively predict healthy coping, mindfulness, coping self-efficacy, and well-being and negatively predict stress and unhealthy coping at the 6-month follow-up and that this would be moderated by sustainability group (i.e., workshop booster sessions, online community drop-ins, digital infographic reminders).

DETAILED DESCRIPTION:
University students face heightened levels of stress and difficulties in coping with daily stressors (American College Health Association, 2023; Ribeiro et al., 2018). The transition to higher education can introduce a variety of stressors such as financial hardships, pressures of novel relationships, and the challenges of unfamiliar social environments, placing students at elevated risk for mental health difficulties (Arnett et al., 2014; Beiter et al., 2015; Ribeiro et al., 2018). Thus, there is a need to provide university students with evidence-based strategies to build their coping and stress management capacity during this exciting but challenging developmental period. As a result, universities are increasingly implementing complementary support services, such as digital self-guided supports (Benjet, 2023; Wang et al., 2023). Digital self-guided resources can be used completely independently (e.g., at the user's own convenience, in terms of time and location of use) and without real-time guidance from a professional or peer (Ahuvia et al., 2024; Edge et al., 2023). These self-guided approaches tend to be less resource-intensive while remaining effective in enhancing student well-being (Amanvermez et al., 2022; Harrer et al., 2019; Oey et al., 2023). Additionally, given university students' reported barriers to accessing mental health services, such as lack of time and a preference for self-management (Benjet, 2023; Dunley & Papadopoulos, 2019; Ebert et al., 2019), digital self-guided resources offer a potential first step for students who are reluctant to engage with traditional approaches to mental health support.

Although digital self-guided resources have been shown to be effective over short periods of time, what is less clear is how to ensure students' long-term use of the strategies being taught in these resources (Harrer et al., 2019; Heber et al., 2017). The majority of studies only examine the short-term effectiveness (i.e., three months or less) of digital self-guided resources (Harrer et al., 2019; Taylor et al., 2024; Wang et al., 2023; Yusufov et al., 2019). However, some studies suggest that users' sustained long-term use of self-guided resources, commonly defined as 3 months or more, is variable and generally low (Fleming et al., 2018; Lattie et al., 2019). In this literature review, the term "resource" is used to define the delivery mechanisms (e.g., mobile apps, infographics, online programs) that provide access to stress management content, while "strategies" refer to the specific coping techniques taught within these resources (e.g., breathing, mindfulness meditation). However, many studies do not differentiate between these terms and will report usage metrics without differentiating between participants' engagement with the resource itself, the strategies included, or both. As such, these terms have been used interchangeably throughout the literature review. Barriers related to long-term use include difficulties remembering to use the strategies and time constraints (Bamber & Schneider, 2022; Kaufman & Nemeroff, 2024; Lyzwinski et al., 2018; Renfrew et al., 2021; Stallman et al., 2020). Such findings highlight a need to expand research in this area by moving away from simply looking at short-term strategy effectiveness towards understanding sustainability approaches that promote long-term strategy use (Gan et al., 2021; Lattie et al., 2019; Taylor et al., 2024).

A common first step in understanding sustained strategy use, defined as ongoing or continued use of the strategies over time, is to consider adherence. Adherence typically refers to the extent to which users follow recommended guidelines for resource use, including the frequency, duration, and program completion (Achilles et al., 2020; Saleem et al., 2021). Measuring adherence is important, as it provides insight into whether students are engaging with interventions as intended (Achilles et al., 2020). However, focusing solely on adherence may not capture the broader and more nuanced patterns of how students continue using specific strategies in their day-to-day lives after initial exposure (Saleem et al., 2021; Taylor et al., 2024; Yusufov et al., 2019). To address this gap, researchers are increasingly exploring the concept of sustained strategy use, which focuses on long-term consistent engagement with specific coping methods beyond the initial intervention period (e.g., Borghouts et al., 2021; Melcher et al., 2022). Sustained strategy use may help students manage stress more effectively by encouraging consistent engagement with healthy coping methods. Particularly when no healthy strategies are perceived as effective or available, individuals remain motivated to alleviate their distress and may instead turn to unhealthy coping strategies; thus, students can be better equipped to manage difficult emotions (Stallman, 2020; Stallman et al., 2020). However, the literature remains unclear on the key areas to support long-term sustained strategy use, especially among university students.

Two key areas that have been suggested to contribute to sustained strategy use are: (1) sustainability supports and (2) the maintenance of behaviour change framework (Alkhaldi et al., 2016; Gan et al., 2021; Kwasnicka et al., 2016). Sustainability supports encompass a variety of approaches aimed at encouraging continued use of wellness strategies. These include providing psychoeducational information on habit formation, sending text or email reminders, and creating accountability groups (Alkhaldi et al., 2016; Gan et al., 2021). On the other hand, maintenance of behaviour change refers to psychological and environmental factors that promote long-term behaviour adoption, such as motivation, self-regulation, habit formation, availability of internal resources, and social/environmental factors (Kwasnicka et al., 2016). Thus, sustainability supports emphasize how to keep students engaged over time, while the maintenance of behaviour change framework focuses on why students continue using strategies in the long term.

The literature outlines a range of diverse sustainability supports, commonly offering information on habit formation (e.g., implementation supports and common barriers to strategy use; Borghouts et al., 2021; Gan et al., 2021; Saleem et al., 2021), fostering community through accountability groups or social support (e.g., peer support; Alkhaldi et al., 2016; Borghouts et al., 2021; Saleem et al., 2021; Vis et al., 2018), and sending text or email reminders (Achilles et al., 2020; Alkhaldi et al., 2016; Saleem et al., 2021). Offering information on habit formation has been suggested as an approach for sustained strategy use by providing psychoeducation and addressing common challenges in developing habits (Borghouts et al., 2021; Gan et al., 2022; Saleem et al., 2021). In university settings, this approach along with wellness services are frequently delivered in the form of workshops (Cho et al., 2024; Yuen et al., 2020), which allow trained facilitators to reach large numbers of students, provide support, and answer questions in real time. Another widely used approach to encourage sustained strategy use is incorporating community-based or peer support components, given the reported influence of social support on engagement (Achilles et al., 2020; Alkhaldi et al., 2016; Saleem et al., 2021). For instance, when participants perceive that an intervention fosters social engagement, whether through facilitator interactions or peer connections, they tend to show higher engagement with the resource and greater use of the strategies offered (Borghouts et al., 2021). Finally, strategy use reminders are also a commonly implemented approach due to their low resource intensity (Borghouts et al., 2021). Reminders have been recommended to support engagement and can be delivered either through SMS/text messages, email, or directly through the resource (i.e., app or gamification software; (Saleem et al., 2021; Zarski et al., 2016). Reminders have been used in several studies to promote strategy use and behaviour change(Clarke et al., 2009; Dryman et al., 2017; Morris et al., 2015; Zarski et al., 2016). Although there is variability in their effectiveness ranging from about 25% to 60%, generally they have been shown to be beneficial (Fry & Neff, 2009; Saleem et al., 2021). It is hypothesized that the variability in effectiveness is due to design and delivery of the interventions rather than the use of reminders themselves. However, to our knowledge, there is no research comparing the effectiveness of these sustainability supports both relative to one another and against an inactive control. As a result, student mental health services are often forced to make decisions without clear data on which approaches are most likely to support sustained strategy use over time.

Another approach to sustaining strategy use involves fostering a behavioural shift (i.e., from non-use or inconsistent use to consistent use of the strategies), thus achieving maintenance of behaviour change. The conceptualization of maintenance of behaviour change as a distinct construct was developed by Kwasnicka et al. (2016) following a review of the literature examining over 100 behaviour change theories and frameworks focusing broadly on health behaviours encompassing both physical and mental health. According to Kwasnicka et al. (2016), the maintenance of behaviour change is underpinned by five interrelated theoretical areas: (1) maintenance motives; (2) self-regulation; (3) habits; (4) internal resources; and (5) environmental/social influences. Maintenance motives refer to various drivers (e.g., behaviour enjoyment, satisfaction with behavioural outcomes, or alignment with the individuals' identity, beliefs and values) that support the ongoing use of the behaviour. Self-regulation refers to the act of consciously managing automatic responses such as behaviours, impulses, desires, or emotions and instead responding in ways that support the desired behaviour. Self-regulation can support an individual in coping with challenges like temptations, setbacks, and relapse (i.e., the risk of returning to the old undesired behaviour). Maintenance of behaviour change is more likely to occur when a habit is formed, which refers to an automatic behaviour that is triggered by contextual cues and develops from consistent self-regulation of the desired behaviour. Ensuring that both psychological and physiological internal resources are plentiful is also an important area of maintenance of behaviour change. When one's resources are depleted, it can be difficult to engage in sustained self-regulation to support maintenance of behaviour change. Finally, maintenance of behaviour change emphasizes that environmental factors and social influences shape behavioural responses and habit formation, especially when social norms support the new desired behaviour. Furthermore, people are more likely to adopt and maintain new behaviours when they feel connected to and supported by a trusted group (Kwasnicka et al., 2016).

Together, these five areas offer a new comprehensive framework for understanding long-term maintenance of behaviour change. Importantly, maintenance of behaviour change provides a distinction between motives that initiate behaviour change and those that sustain it. Despite the framework's conceptual strengths and use in the health context, its application within mental health remains underexplored. To our knowledge, the relationship between maintenance of behaviour change and wellness outcomes and the comparative impact of sustainability approaches has yet to be explored.

Building on these insights and addressing the noted gaps, Click or tap here to enter text.Click or tap here to enter text.Click or tap here to enter text.the current study evaluates which types of sustainability support best promote wellness outcomes, sustained strategy use, and maintenance of behaviour change as well as identifying which sustainability support students find most acceptable. Moreover, this study examines whether maintenance of behaviour change may predict long-term wellness benefits and whether this relationship is strengthened or weakened based on sustainability group.

Therefore, the overarching objective of the current study is to evaluate the effectiveness, acceptability, strategy use, and maintenance of behaviour change of different stress management sustainability groups. Furthermore, the study aims to examine how these sustainability groups and maintenance of behaviour change may impact student wellness in the long term. Specifically, objective 1 sought to compare three commonly employed approaches for sustainability of stress management strategy use (workshop booster sessions, online community drop-ins, digital infographic reminders) and an inactive control group (no support) in terms of their (1.1) effectiveness on wellness outcomes (i.e., stress, healthy and unhealthy coping capacity, mindfulness, coping self-efficacy, and well-being), (1.2) acceptability, (1.3) strategy use, and (1.4) maintenance of behaviour change over time. It was hypothesized that the community drop-in sustainability group would have greater effectiveness, strategy use, and maintenance of behaviour change compared to the other sustainability groups and inactive control. This hypothesis aligns with the literature across both sustainability supports and maintenance of behaviour change-related indices, suggesting that social support is a key element to sustained strategy use (Borghouts et al., 2021; Kelders et al., 2012; Kwasnicka et al., 2016). No specific hypothesis was made for which sustainability approach would be rated as most (H1.2) acceptable given this is a novel area of research.

Objective 2 sought to examine (2.1) whether maintenance of behaviour change at post (T2) predicted wellness outcomes (i.e., stress, healthy and unhealthy coping capacity, mindfulness, coping self-efficacy, and well-being) at 6-month follow-up (T4), and whether this relationship was differentially moderated by sustainability group. It was hypothesized (H2.1) that maintenance of behaviour change at post would positively predict healthy coping, mindfulness, coping self-efficacy, and well-being and negatively predict stress and unhealthy coping at the 6-month follow-up and that this would be moderated by sustainability group (i.e., workshop booster sessions, online community drop-ins, digital infographic reminders).

Method: Phase 1 focused on the development of the stress management resource. All participants received the same interactive stress management infographic (i.e., with embedded links for strategy practice), which was evaluated in a previous study (see Bastien et al., under review). This brief three-page interactive infographic was created following a critical review of the literature identifying key areas for coping with stress, specifically: (a) being in the moment; (b) enhancing positive emotions through mindfulness and gratitude; (c) practicing self-compassion; and (d) seeking social support. The brief interactive infographic contained both psychoeducational content and strategy introduction as well as embedded skills-based practice of stress management strategies tailored for university students.

Subsequently, in Phase 2, different sustainability approaches were developed to ensure equivalent content across: (a) psychoeducation on habit formation and maintenance of behaviour change; and (b) embedded skills-based practice of habit formation. Mirroring Phase 1, content for the sustainability groups was developed following a critical review of the literature on habit formation and maintenance of behaviour change (e.g., Achilles et al., 2020; Alkhaldi et al., 2016; Borghouts et al., 2021; Kwasnicka et al., 2016; Saleem et al., 2021; Zhu et al., 2024). Themes addressed in the sustainability approaches included: (a) understanding values; (b) goal setting; (c) planning for challenges; (d) awareness of resources; (e) facing setbacks; (f) building a community of practice; and (g) general tips for getting started. The sustainability groups consisted of:

* Workshop Boosters: Two 45-minute online workshop boosters presented about two months apart, led by two trained undergraduate peer facilitators with 10 to 20 participants per session.
* Community Drop-in Sessions: Five monthly 20-minute online community drop-in sessions held over a five-month period, led by the same facilitators with 10-15 participants.
* Infographic Reminders: Ten brief digital infographic reminders (one to two pages each) emailed to students once every two weeks over a five-month period.

Following each workshop and community drop-in session, students were emailed a brief one-page resource sheet with links to the strategies for habit formation presented in the session. All sustainability groups were identical in the content provided but differed in terms of the modality in which it was presented. The inactive control group did not receive any sustainability support throughout the study (they only had access to the initial stress management resource), but they received access to all the sustainability materials at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* University students

Exclusion Criteria:

-

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 331 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Change in stress | baseline, 1-month , 3-month, and 6-month follow-up
  The Perceived Stress Scale (PSS) is a widely used self-report measure of individuals' perception of stress. This measure contains 10 items in which participants indicate their experience of stress on a 5-point Likert scale (0 = never to 4 = very often). Items were adapted to reflect experiences during the past week and include statements such as "In the past week, how often have you felt difficulties were piling up so high that you could not overcome them?" Ratings were averaged across items such that higher scores represented greater perceived stress. The PSS has good reliability (Cronbach's α = .89), construct validity, and predictive validity with reports of psychological and physical symptoms.

SECONDARY OUTCOMES:
Group differences on satisfaction | 1-month , 3-month, and 6-month follow-up
  The Response to Training is a researcher-developed questionnaire assessing participants' satisfaction with the sustainability intervention content and delivery. The questions were delivered according to the three levels of Kirkpatrick's New World Model (Kirkpatrick & Kirkpatrick, 2016) as follows: (1) student viewers' response (i.e., satisfaction, engagement, relevance); (2) learning (i.e., knowledge, skills, attitude, confidence, commitment); (3) use of skills (i.e., willingness to use, frequency of use). All items are scored on a 6-point Likert-scales except for the strategy use item described below, where higher scores represent a better response to training. Sample items include "I would recommend the sustainability support to other university students" or "I am planning to use the strategies in the future..."
Change in coping capacity | baseline, 1-month , 3-month, and 6-month follow-up
  The Coping Index (CI; (Stallman, 2017), a 20-item measure of engagement with healthy and unhealthy coping strategies that are aligned with the health theory of coping framework (Stallman, 2020). The measure consists of items that list common healthy and unhealthy coping behaviours such as 'talk things over with family or friends', 'do relaxing activities', or 'have negative self-talk'. Participants are asked to indicate how often they engage in each behaviour listed when they feel stressed or distressed on a 4-point Likert scale (0 = I don't do this at all to 3 = I do this most of the time). This measure has been found to have satisfactory test-retest reliability with alpha = 0.71 (Stallman, 2019).
Change in mindfulness | baseline, 1-month , 3-month, and 6-month follow-up
  The Five Facets of Mindfulness Questionnaire short form (FFMQ-15; (Baer et al., 2006, 2008) which is a 15-item self-report measure consisting of five subscales each assessing a specific facet of dispositional mindfulness: acting with awareness, describing, observing, non-reactivity, and non-judgmental acceptance. Items include "I'm good at finding words to describe my feelings" and "When I have distressing thoughts or images, I am able just to notice them without reacting". Participants rate their responses on a 5-point Likert scale (1 = never or very rarely true to 5 = very often or always true). The FFMQ-15 has good internal consistency with Cronbach alphas ranging from .64 to .83, as well as convergent validity (Gu et al., 2016). Higher scores on the FFMQ-15 represent higher mindfulness.
Change in coping self-efficacy | baseline, 1-month , 3-month, and 6-month follow-up
  The Coping Self-Efficacy Scale (CSES; Chesney et al., 2006) which is a measure of one's confidence in effectively engaging in coping behaviors in the face of challenges. This measure contains 26 items in which participants indicate confidence in their coping strategies when it comes to handling challenges and stressors on an 11-point Likert scale (0 = cannot do at all to 10 = certain can do). The CSES states, "When things aren't going well for you, or when you're having problems, how confident or certain are you that you can do the following:" and include statements such as "find solutions to your most difficult problems" and "see things from the other person's point of view during a heated argument." Higher scores on the CSES represent higher coping-self efficacy.
Change in well-being | baseline, 1-month , 3-month, and 6-month follow-up
  The Warwick-Edinburg Mental Well-Being Scale (WEMWBS; Tennant et al., 2007), which is a measure of positive mental health and consists of 14 positively worded items. Participants are asked to rate statements such as "I've been feeling good about yourself" on a 5-point Likert scale according to their experience over the past 2 weeks (1= none of the time; 5= all of the time). The WEMWBS has demonstrated good internal consistency in student (α = .89) and general population samples (α = .91) and was found to be psychometrically robust in validation studies (Stewart-Brown et al., 2011; Tennant et al., 2007).
Change in maintenance of behaviour change | 1-month , 3-month, and 6-month follow-up
  Maintenance of Behaviour Change is a 17-item researcher-developed measure based on Kwasnicka et al.'s (2016) theoretical framework for maintenance of behaviour change. The measure assesses an individual's ability to adopt and maintain long-term stress management strategy use (i.e., behaviour change). Specifically, items were developed from each of Kwasnicka et al.'s (2016) five main areas for maintenance of behaviour change which include: (1) maintenance motives; (2) self-regulation; (3) habits; (4) internal resources; and (5) environmental/social influences. In the present study, internal consistency for the maintenance of behaviour change measure was good (α = .89, .91, and .91 at T2, T3, and T4, respectively). The sum score of the item was used with a maximum score of 85. Higher scores on the measure indicate better maintenance of behaviour change.
Stress management strategy use | 1-month , 3-month, and 6-month follow-up
  Strategy use was measured using a researcher-designed item developed from the third level of Kirkpatrick's New World Model (Kirkpatrick & Kirkpatrick, 2016) assessing use of skill. Using a 4-point Likert scale (never, rarely, sometimes, frequently, everyday), participants were asked, "Over the past two weeks, how often did you use the strategies presented in the infographic stress management resource?" Higher scores indicate greater use of the stress management strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Heath, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor ME, Liu M, Abelson S, Eisenberg D, Lipson SK, Schueller SM. The Reach, Effectiveness, Adoption, Implementation, and Maintenance of Digital Mental Health Interventions for College Students: A Systematic Review. Curr Psychiatry Rep. 2024 Dec;26(12):683-693. doi: 10.1007/s11920-024-01545-w. Epub 2024 Oct 11. PMID 39392547
- [Background] Saleem M, Kuhne L, De Santis KK, Christianson L, Brand T, Busse H. Understanding Engagement Strategies in Digital Interventions for Mental Health Promotion: Scoping Review. JMIR Ment Health. 2021 Dec 20;8(12):e30000. doi: 10.2196/30000. PMID 34931995
- [Background] Oey LT, McDonald S, McGrath L, Dear BF, Wootton BM. Guided versus self-guided internet delivered cognitive behavioural therapy for diagnosed anxiety and related disorders: a preliminary meta-analysis. Cogn Behav Ther. 2023 Nov;52(6):654-671. doi: 10.1080/16506073.2023.2250073. Epub 2023 Sep 1. PMID 37655553
- [Background] Lattie EG, Adkins EC, Winquist N, Stiles-Shields C, Wafford QE, Graham AK. Digital Mental Health Interventions for Depression, Anxiety, and Enhancement of Psychological Well-Being Among College Students: Systematic Review. J Med Internet Res. 2019 Jul 22;21(7):e12869. doi: 10.2196/12869. PMID 31333198
- [Background] Heber E, Ebert DD, Lehr D, Cuijpers P, Berking M, Nobis S, Riper H. The Benefit of Web- and Computer-Based Interventions for Stress: A Systematic Review and Meta-Analysis. J Med Internet Res. 2017 Feb 17;19(2):e32. doi: 10.2196/jmir.5774. PMID 28213341
- [Background] Harrer M, Adam SH, Baumeister H, Cuijpers P, Karyotaki E, Auerbach RP, Kessler RC, Bruffaerts R, Berking M, Ebert DD. Internet interventions for mental health in university students: A systematic review and meta-analysis. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1759. doi: 10.1002/mpr.1759. Epub 2018 Dec 26. PMID 30585363
- [Background] Fleming T, Bavin L, Lucassen M, Stasiak K, Hopkins S, Merry S. Beyond the Trial: Systematic Review of Real-World Uptake and Engagement With Digital Self-Help Interventions for Depression, Low Mood, or Anxiety. J Med Internet Res. 2018 Jun 6;20(6):e199. doi: 10.2196/jmir.9275. PMID 29875089
- [Background] Edge D, Watkins ER, Limond J, Mugadza J. The efficacy of self-guided internet and mobile-based interventions for preventing anxiety and depression - A systematic review and meta-analysis. Behav Res Ther. 2023 May;164:104292. doi: 10.1016/j.brat.2023.104292. Epub 2023 Mar 22. PMID 37003138
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Arnett JJ, Zukauskiene R, Sugimura K. The new life stage of emerging adulthood at ages 18-29 years: implications for mental health. Lancet Psychiatry. 2014 Dec;1(7):569-76. doi: 10.1016/S2215-0366(14)00080-7. Epub 2014 Dec 3. PMID 26361316
- [Background] Amanvermez Y, Zhao R, Cuijpers P, de Wit LM, Ebert DD, Kessler RC, Bruffaerts R, Karyotaki E. Effects of self-guided stress management interventions in college students: A systematic review and meta-analysis. Internet Interv. 2022 Feb 12;28:100503. doi: 10.1016/j.invent.2022.100503. eCollection 2022 Apr. PMID 35242591
- [Background] Achilles MR, Anderson M, Li SH, Subotic-Kerry M, Parker B, O'Dea B. Adherence to e-mental health among youth: Considerations for intervention development and research design. Digit Health. 2020 May 21;6:2055207620926064. doi: 10.1177/2055207620926064. eCollection 2020 Jan-Dec. PMID 32547775